CLINICAL TRIAL: NCT04642326
Title: Prospective, Parallel, Multicenter Randomized Controlled Study Investigating the Effects of UVC Beam and Laser Beam Therapy According to Standard Therapy in Patients With Covid-19 Diagnosis
Brief Title: Study Investigating the Effects of UVC Beam and Laser Beam Therapy According to Standard Therapy in Patients With Covid-19 Diagnosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RD Global Araştirma Geliştirme Sağlik Ilaç Inşaat Yatirimlari A.Ş. (Industry)
Responsible Party: Principal Investigator, Hikmet Selçuk Gedik, Cardiovascular Surgeon, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD2020/001
Record Dates: First submitted 2020-11-16; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Prospective, Parallel, Multicenter Randomized Controlled Study Investigating
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group: experimental - UVC Therapy applied (Experimental): Test: Antiviral + Antimalarial + Antibiotic Treatment + UVC Therapy
  Interventions: Device: Test Group: experimental - UVC Therapy applied
- Control Group (No Intervention): Control: Antiviral + Antimalarial + Antibiotic Treatment

INTERVENTIONS:
Device: Test Group: experimental - UVC Therapy applied — in addition to traditional drug therapy, apply a surgical treatment procedures with using special UVC device.(Antiviral + Antimalarial + Antibiotic Treatment + UVC Therapy)
  Other Names: of Turkish Beam-Selective UV Device Model Number: 1007-001
  Arms: Test Group: experimental - UVC Therapy applied

SUMMARY:
Clinical research study that evaluates the effect of Turkish Beam-Selective UV developed by RD GLOBAL ARAŞTIRMA GELİŞTİRME SAĞLIK İLAÇ İNŞAAT YATIRIMLARI A.Ş. use into Intravascular, Intrapulmonary, Intratracial, Intrarespiratory area. Bacteria, Fungal and Virus-based pathogens systematically to collect and evaluate specific clinical performance and safety data.

This Clinical Research aims to investigate the effectiveness of the treatment group and control group mortality rates, intensive care hospitalization times, monitoring the virus load by PCR, and the treatment effectiveness of UVC application.

This Clinical Research covers determining the treatment effectiveness and reliability of UVC application to patient groups, the details of which are determined in the protocol.

DETAILED DESCRIPTION:
DESIGN

Prospective, parallel, multicentre, randomized controlled study Ages between 40 and 75 years of age and positive symptoms such as fever, malaise, cough, and shortness of breath, or positive atypical pneumonia in CT findings or COVID-19 (SARS-CoV-2) test In the intensive care unit, which is accepted as COVID 19 infection and has been treated, patients will be treated with UVC radiation and laser beam treatment according to IKU principles in addition to Antimalarial therapy + Antiviral therapy + Anitibiotic therapy. Standard treatment consisting of Antimalarial therapy + Antiviral therapy + Antibiotic therapy will be applied to the control group. The dosage of the standard treatment consisting of antimalarial therapy + Antiviral therapy + Anitibiotic therapy, the number of days of treatment, and its active ingredient are indicated in the table.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory rate ≥ 30
* Dyspnea and breathing difficulties findings
* Cases with oxygen saturation below 90% despite nasal oxygen support of 5 liters / minute and above
* Cases with partial oxygen pressure below 70 mmHg despite nasal oxygen support of 5 liters / minute and above
* PaO2 / FiO2 <300 Lactate> 4 mmol / L Bilateral infiltrations or multi-lobar involvement on chest x-ray or tomography
* Hypotension (systolic blood pressure <90 mmHg,> 40 mmHg drop from usual SKB, mean arterial pressure <65 mmHg)
* Skin perfusion disorder Organ dysfunction such as kidney function test, liver function test disorder, thrombocytopenia, confusion Presence of immunosuppressive disease- Presence of uncontrolled comorbidity with more than one feature
* Troponin height, arrhythmia
* COVID 19 Test positivity

Exclusion Criteria:

* Under 40 years old
* Pregnant women and those with suspected pregnancy
* Those with a history of anaphylaxis
* Those with known DNA repair deficiencies:
* Those diagnosed with mental disorder,
* puerperant women and lactating women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-05-04 (Estimated)

PRIMARY OUTCOMES:
PCR Sampling | up to 15 days
  viral load measurement due to covid 19,
Blood Tests | up to 15 days
  Change from reference range in blood urea (mg/dL)
Blood Tests | up to 15 days
  Change from reference range in blood Creatinine (mg/dL)
Blood Tests | up to 15 days
  Change from reference range in blood AST,ALT (U/L)
Blood Tests | up to 15 days
  Change from reference range in Complete blood count (sodium, potassium mol/L)
Blood Tests | up to 15 days
  Change from reference range in Complete blood count (total bilirubin mg/dL)
Blood Tests | up to 15 days
  Change from reference range in Complete blood CRP (mg/L)
Blood Tests | up to 15 days
  Change from reference range in Complete blood creatine kinase (IU/L)
Blood Tests | up to 15 days
  Change from reference range in Complete blood LDH (U/L)
Blood Tests | up to 15 days
  Change from reference range in Complete blood APTT (sec)
Blood Tests | up to 15 days
  Change from reference range in Complete blood D-Dimer (ng/ml)
Blood Tests | up to 15 days
  Change from reference range in Complete blood Ferritin (ug/L)
Radiological Imaging | up to 15 days
  Radiological findings: Consolidation, ground glass appearance and reticulo-nodular opacity appearance in lung CT.
Radiological Imaging | up to 15 days
  Radiological findings: reticulo-nodular opacity appearance in lung CT.
Radiological Imaging | up to 15 days
  Radiological findings: ground glass appearance in lung CT.
Radiological Imaging | up to 15 days
  Radiological findings: Consolidation in lung CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Diyarbakır SBÜ Gazi Yaşargil Eğitim Ve Araştırma Hastanesi, Diyarbakır, Kayapınar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
During or when the study ends, the data will be shared for scientific publication.

REFERENCES:
- [Background] Kim S, Kim J, Lim W, Jeon S, Kim O, Koh JT, Kim CS, Choi H, Kim O. In vitro bactericidal effects of 625, 525, and 425 nm wavelength (red, green, and blue) light-emitting diode irradiation. Photomed Laser Surg. 2013 Nov;31(11):554-62. doi: 10.1089/pho.2012.3343. Epub 2013 Oct 19. PMID 24138193
- [Background] Cheng VC, Lau SK, Woo PC, Yuen KY. Severe acute respiratory syndrome coronavirus as an agent of emerging and reemerging infection. Clin Microbiol Rev. 2007 Oct;20(4):660-94. doi: 10.1128/CMR.00023-07. PMID 17934078
- [Result] Yin R, Dai T, Avci P, Jorge AE, de Melo WC, Vecchio D, Huang YY, Gupta A, Hamblin MR. Light based anti-infectives: ultraviolet C irradiation, photodynamic therapy, blue light, and beyond. Curr Opin Pharmacol. 2013 Oct;13(5):731-62. doi: 10.1016/j.coph.2013.08.009. Epub 2013 Sep 20. PMID 24060701
- [Result] Mohr H, Steil L, Gravemann U, Thiele T, Hammer E, Greinacher A, Muller TH, Volker U. A novel approach to pathogen reduction in platelet concentrates using short-wave ultraviolet light. Transfusion. 2009 Dec;49(12):2612-24. doi: 10.1111/j.1537-2995.2009.02334.x. Epub 2009 Aug 4. PMID 19682340
- [Result] Galasso M, Feld JJ, Watanabe Y, Pipkin M, Summers C, Ali A, Qaqish R, Chen M, Ribeiro RVP, Ramadan K, Pires L, Bagnato VS, Kurachi C, Cherepanov V, Moonen G, Gazzalle A, Waddell TK, Liu M, Keshavjee S, Wilson BC, Humar A, Cypel M. Inactivating hepatitis C virus in donor lungs using light therapies during normothermic ex vivo lung perfusion. Nat Commun. 2019 Jan 29;10(1):481. doi: 10.1038/s41467-018-08261-z. PMID 30696822
- [Result] Eickmann M, Gravemann U, Handke W, Tolksdorf F, Reichenberg S, Muller TH, Seltsam A. Inactivation of three emerging viruses - severe acute respiratory syndrome coronavirus, Crimean-Congo haemorrhagic fever virus and Nipah virus - in platelet concentrates by ultraviolet C light and in plasma by methylene blue plus visible light. Vox Sang. 2020 Apr;115(3):146-151. doi: 10.1111/vox.12888. Epub 2020 Jan 12. PMID 31930543
- [Result] Dai T, Kharkwal GB, Zhao J, St Denis TG, Wu Q, Xia Y, Huang L, Sharma SK, d'Enfert C, Hamblin MR. Ultraviolet-C light for treatment of Candida albicans burn infection in mice. Photochem Photobiol. 2011 Mar-Apr;87(2):342-9. doi: 10.1111/j.1751-1097.2011.00886.x. Epub 2011 Feb 10. PMID 21208209
- [Result] Cypel M, Feld JJ, Galasso M, Pinto Ribeiro RV, Marks N, Kuczynski M, Kumar D, Bahinskaya I, Bagnato VS, Kurachi C, Slutsky AS, Yeung JC, Donahoe L, de Perrot M, Yasufuku K, Pierre A, Binnie M, Chaparro C, Martinu T, Chen M, Tikkanen J, Chow CW, Sidhu A, Waddell TK, Keshavjee S, Singer LG, Humar A. Prevention of viral transmission during lung transplantation with hepatitis C-viraemic donors: an open-label, single-centre, pilot trial. Lancet Respir Med. 2020 Feb;8(2):192-201. doi: 10.1016/S2213-2600(19)30268-1. Epub 2019 Oct 9. PMID 31606437
- [Result] Bak J, Jorgensen TM, Helfmann J, Gravemann U, Vorontsova I. Potential in vivo UVC disinfection of catheter lumens: estimation of the doses received by the blood flow outside the catheter tip hole. Photochem Photobiol. 2011 Mar-Apr;87(2):350-6. doi: 10.1111/j.1751-1097.2011.00887.x. Epub 2011 Jan 31. PMID 21208210
- [Result] Ultroviolet,C lrrodiation for Prevention of Centrol Venous Cotheter-reloted · lnfections: An in Vitro Study,Tianhong Dai 1,2, George P. Tegos 1,2§, Tyler G. St. Denis l ,3, Don Anderson4,. Ed SinofskyS ond Michael R. Homblin* l ,2,6, Received 11 Moy 201 O, accepted 8 September 201 o; DOi: l 0.1111/ j.1751-1097.2010.00819 .x
- [Result] Pathogen inactivation method using ultraviolet C light. Journal of Transfusion Medicine, 12(3), 83-87.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT04642326/Prot_SAP_000.pdf